CLINICAL TRIAL: NCT06537544
Title: Comparison of Comprehensive Rehabilitation Program and Conventional Pelvic Floor Training in Women With Stress Urinary Incontinence
Brief Title: Comparison of Comprehensive Rehab Program and Pelvic Floor Training in Women With Stress Urinary Incontinence
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Shahzadi Safoora Shamail
Record Dates: First submitted 2024-07-27; First posted 2024-08-05 (Actual); Last update posted 2025-03-05 (Actual); Status verified 2025-03

CONDITIONS: Stress Urinary Incontinence
MeSH Terms: conditions — Urinary Incontinence, Stress

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Conventional Pelvic Floor Training (Active Comparator): This group will receive pelvic floor muscle training exercises in supine, sitting , kneeling and standing position with gradual increase in frequency, dosage and duration of exercises.
  Interventions: Other: Conventional Pelvic Floor Training
- Comprehensive Rehabilitation Program (Experimental): This group will receive Core Strengthening Exercises, Breathing Exercises and education along with Pelvic Floor Muscle Strengthening Exercises
  Interventions: Other: Comprehensive Rehabilitation Program

INTERVENTIONS:
Other: Comprehensive Rehabilitation Program — Pelvic Floor Muscle Strengthening Exercises Core Strengthening Exercises Breathing Exercises Patient education about bladder diary Postural education
  Arms: Comprehensive Rehabilitation Program
Other: Conventional Pelvic Floor Training — Kegels exercises in different body positions
  Arms: Conventional Pelvic Floor Training

SUMMARY:
The goal of this clinical trial is to compare a comprehensive rehabilitation program and a conventional pelvic floor training program in women with stress urinary incontinence,to compare the effects of comprehensive rehabilitation program and conventional pelvic floor training on the severity of SUI, on the strength of pelvic floor muscle and on quality of life in women with SUI. Following the randomization into either the conventional pelvic floor training or comprehensive rehabilitation program group, participants will receive their assigned interventions of three weekly sessions for eight weeks.

DETAILED DESCRIPTION:
The proposed study comparing the effects of conventional pelvic floor training versus a comprehensive rehabilitation program on stress urinary incontinence (SUI) among perimenopausal women holds significant rationale and importance. Given the prevalence and impact of SUI on the quality of life of perimenopausal women, investigating the comparative efficacy of these interventions is crucial for informing evidence-based clinical practice. The study aims to provide insights into the most effective management strategies for SUI in this population, potentially leading to improved treatment outcomes, enhanced quality of life, and reduced healthcare burden associated with this common condition. By addressing this research gap, the study has the potential to significantly benefit both individual patients and the broader healthcare system.

This will be a randomized controlled trial. Non probability sampling technique will be used.The data collection procedure begins with the recruitment phase, potential participants meeting the study's criteria will be identified and provided with detailed information about the research aims and procedures. Once recruited, participants will undergo a screening process to confirm their eligibility, including assessments such as medical history reviews and diagnostic tests. After obtaining informed consent, baseline assessments will be conducted to establish the participants' initial status regarding urinary symptoms and quality of life. Following randomization into either the conventional pelvic floor training or comprehensive rehabilitation program group, participants will receive their assigned interventions of three weekly sessions for eight weeks.

ELIGIBILITY:
Inclusion Criteria:

* Perimenopausal and post-menopausal women
* Age 40-60 years
* Medically diagnosed patients of stress urinary incontinence

Exclusion Criteria:

* History of pelvic surgery within the past six months.
* Current urinary tract infections or other active urinary tract disorders.
* Neurological conditions affecting bladder control.
* Inability to participate in the prescribed intervention due to physical or cognitive limitations.
* Participation in other pelvic floor rehabilitation programs concurrently or previously within the last 6 months.

Ages: 40 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 62 (Actual)
Dates: Start 2024-08-01 (Actual); Primary Completion 2025-01-10 (Actual); Study Completion 2025-01-10 (Actual)

PRIMARY OUTCOMES:
Severity of stress urinary incontinence | Changes from Baseline to 8 weeks
  To compare the effects of comprehensive rehabilitation program and conventional pelvic floor training on the severity of stress urinary incontinence

SECONDARY OUTCOMES:
Strength of pelvic floor muscle | Changes from Baseline to 8 weeks
  To compare the effects of comprehensive rehabilitation program and conventional pelvic floor training on the strength of pelvic floor muscle
Quality of life in women with stress urinary incontinence | Changes from Baseline to 8 weeks
  To compare the effects of comprehensive rehabilitation program and conventional pelvic floor training on quality of life in women with stress urinary incontinence

CONTACTS AND LOCATIONS:
Overall Officials: Huma Riaz, PhD, Study Chair — Riphah International University, Islamabad, Pakistan; Shahzadi Safoora Shamail, DPT, Principal Investigator — Riphah International University, Islamabad, Pakistan
Locations (1):
- King Abdullah Teaching Hospital, Mansehra, KPK, Pakistan

IPD SHARING:
Plan to Share IPD: No